CLINICAL TRIAL: NCT00006308
Title: Observational Cohort Study of Sodium, Weight and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy Cook, ScD, Professor, Brigham and Women's Hospital
Other Study IDs: 916; R01HL057915 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate cardiovascular events among individuals with low sodium intake or large weight changes in a prospective observational follow-up of subjects from the Trials of Hypertension Prevention (TOHP) study.

DETAILED DESCRIPTION:
BACKGROUND:

Sodium reduction and weight loss lead to decreased blood pressure (BP). Among hypertensives, BP lowering leads to decreased risk of MI, stroke, and cardiovascular death. Nonetheless, concerns have been raised about increased numbers of cardiovascular events among individuals with low sodium intake or large weight changes.

DESIGN NARRATIVE:

The prospective observational follow-up of the Trials of Hypertension Prevention (TOHP) includes cardiovascular events among the 4, 507 surviving participants from the ten clinical centers involved in Phases I and II of TOHP. Phase I was a randomized trial of the effects of non- pharmacologic interventions, including sodium reduction and weight loss, on BP over 18 months of follow-up with 2,182 participants. Phase II examined the effects of sodium reduction and weight loss on BP over a longer 36-month period in a randomized 2X2 factorial design with 2,382 participants. During follow-up in Phases I and II of TOHP, several measures of both weight and sodium excretion were carefully obtained on all participants. The prospective observational follow-up specifically examines whether these values, with an emphasis on average level of sodium excretion and weight changes are predictive of later cardiovascular disease. The follow-up is conducted centrally by mail from the Division of Preventive Medicine, which served as the Coordinating Center for Phases I and II, and which has been very successful in conducting such large-scale studies by mail. Information on cardiovascular events subsequent to the trial periods is collected through June, 2003, representing an average follow-up of approximately fourteen years from the end of Phase I and eight years from the end of Phase II. This cohort provides a unique resource to address the impact in a normotensive population of salt restriction and weight change on subsequent cardiovascular events.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Cook, ScD, Principal Investigator — Brigham and Women's Hospital